CLINICAL TRIAL: NCT07327723
Title: The Effects of Repetitive Peripheral Magnetic Stimulation on Clinical and Electrophysiological Parameters in Patients With Carpal Tunnel Syndrome: A Double-Blind, Randomized, Sham-Controlled Trial
Brief Title: Effects of Repetitive Peripheral Magnetic Stimulation(rPMS) on CTS(Carpal Tunnel Syndrome)
Acronym: rPMS CTS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Seçilay Güneş, Associated Professor, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-480-25; TTU-2025-4307 (Other Grant/Funding Number: Ankara University Scientific Research Project Coordination)
Record Dates: First submitted 2025-11-17; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: Carpal Tunnel Syndrome; Repetitive Peripheral Magnetic Stimulation; electrodiagnosis; ultrasound; functional status
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: A Double-Blind, Randomized, Sham-Controlled Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rPMS group (Active Comparator): All patients will be instructed in tendon and nerve gliding exercises by a physiotherapist. In addition to these exercises, the treatment group will undergo repetitive peripheral magnetic stimulation (rPMS) therapy three times per week for two consecutive weeks, for a total of six sessions. Each session will last 10 minutes
  Interventions: Device: rPMS group
- sham- rPMS group (Sham Comparator): All patients will be instructed in tendon and nerve gliding exercises by a physiotherapist. In addition to these exercises, the sham-rPMS group will receive sham repetitive peripheral magnetic stimulation (rPMS) therapy, three times per week for two weeks, totaling six sessions. Each session will last 10 minutes. Patients will be positioned identically, and the device will be placed in the same position but not activated. Instead, previously recorded operational sounds of the device will be played back during the same duration to simulate the treatment experience.
  Interventions: Device: sham-rPMS

INTERVENTIONS:
Device: rPMS group — All patients will be instructed in tendon and nerve gliding exercises by a physiotherapist. In addition to these exercises, the treatment group will undergo repetitive peripheral magnetic stimulation (rPMS) therapy three times per week for two consecutive weeks, for a total of six sessions. Each session will last 10 minutes. The rPMS treatment will be administered using the BTL-6000 Super Inductive System Elite device. From the device interface, the "wrist/hand" region will be selected, and the "carpal tunnel syndrome" protocol pre-programmed for this region will be applied.
  During the procedure, patients will be instructed to lie supine or sit in a relaxed position to ensure complete muscle relaxation in the arm. The applicator will be positioned on the volar aspect of the wrist, aligned with the carpal tunnel, as close to the skin as possible.
  The frequency will be set between 5-50 Hz, and intensity will be adjusted to elicit visibly observable muscle contractions.
  Arms: rPMS group
Device: sham-rPMS — In the sham group, patients will be positioned identically, and the device will be placed in the same position but not activated. Instead, previously recorded operational sounds of the device will be played back during the same duration to simulate the treatment experience.
  All participants will be closely monitored throughout the treatment period
  Arms: sham- rPMS group

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common entrapment neuropathy, resulting from compression of the median nerve at the wrist. It is particularly common in middle-aged women. In the early stages, these patients frequently experience pain and numbness in the hand, especially in the first three fingers, and paresthesias, which often worsen at night. As the disease progresses, muscle weakness and atrophy of the thenar muscles can occur, severely impacting patients' daily activities and functionality. Clinical evaluation and patient complaints are crucial for diagnosis. Electrophysiological assessment tools such as nerve conduction studies and electromyography (EMG) are highly sensitive and considered the gold standard for confirming the diagnosis, assessing nerve damage, and determining the severity of this damage. In addition to electrophysiological assessment, ultrasonographic evaluation offers an important opportunity to observe structural changes in the median nerve associated with CTS.

In cases of mild to moderate CTS, nonsurgical treatments are the primary options for reducing symptoms; splinting, tendon-nerve gliding exercises, and physical therapy modalities are commonly preferred. Repetitive peripheral magnetic stimulation (rPMS) is a non-invasive method that can be applied to various tissues, such as spinal nerves, peripheral nerves, or muscles, and is used to reduce pain and improve motor function. While its potential benefits for many neurological diseases and musculoskeletal problems have been demonstrated in recent years, there are limited studies on the effectiveness of rPMS in patients with CTS. The primary objective of this study is to evaluate the effectiveness of rPMS on pain in individuals diagnosed with mild to moderate CTS. Secondarily, the effects of rPMS on symptom severity, functional status, nerve conduction parameters, and median nerve ultrasonographic findings will be analyzed. The findings of our study suggest that objective evaluation of rPMS treatment will contribute to supporting the clinical practice of this treatment option in patients with CTS with more comprehensive data.

DETAILED DESCRIPTION:
This study is designed as a prospective, randomized, sham-controlled, double-blind, experimental study. It was approved by the Ethics Committee of Ankara University, Faculty of Medicine, and will be conducted in accordance with the Declaration of Helsinki. The study will be conducted at the Department of Physical Medicine and Rehabilitation, Ankara University Faculty of Medicine Hospital. Eligible participants who are over 18 years of age, have provided informed consent, and have clinical symptoms and physical examination findings consistent with carpal tunnel syndrome (CTS), along with electrodiagnostic confirmation of mild to moderate CTS, will be enrolled. Participants will randomly be assigned to two groups: a treatment group and a sham group. Randomization will be performed using the Random Allocation Software (RAS) program. All patients will be instructed in tendon and nerve gliding exercises by a physiotherapist. In addition to these exercises, the treatment group will undergo repetitive peripheral magnetic stimulation (rPMS) therapy three times per week for two consecutive weeks, for a total of six sessions. Each session will last 10 minutes. rPMS will be applied by a physiotherapist who is blinded to the participants' diagnoses and outcome evaluations. All participants will be carefully monitored throughout the intervention period. Assessments will be conducted at three time points: baseline, three weeks after the final treatment session, and six weeks post-treatment. Participants will be assessed by Dr. Sema Köylü Dağ, who will be blinded to patient group allocation and diagnosis, using the case report form. In line with this form, sociodemographic data, including age, sex, height, weight, body mass index (BMI), marital status, educational level, occupation, and contact information, will be recorded, along with medical history, symptom duration, smoking status, dominant hand, and affected hand. Assessments will include the Visual Analog Scale (VAS), grip and pinch strength measurements (kg), the Boston Carpal Tunnel Questionnaire (BCTQ), the Short Form-36 Health Survey (SF-36), electrophysiological evaluation of the median nerve, and ultrasonographic cross-sectional area measurement (mm²) of the median nerve.

Statistical Analysis Sample size was calculated based on the primary endpoint: detecting a clinically meaningful difference in Visual Analog Scale (VAS) scores between the two groups, with a mean effect size of 1.4. Assuming a significance level of α = 0.05 and power = 0.95, the required sample size was calculated as 15 patients per group (30 patients in total). Calculations were performed using the GPower 3.1 software. Considering possible dropouts, the plan is to recruit 20 participants per group, totaling 40 patients.

Descriptive statistics will be presented as mean ± standard deviation, median (minimum-maximum), and frequency (percentage).

For between-group comparisons, Student's t-test and chi-square test will be used.

For within-group comparisons, repeated measures ANOVA or the Friedman test will be employed.

Correlations between variables will be analyzed using Pearson correlation coefficient.

A p-value < 0.05 will be considered statistically significant

ELIGIBILITY:
Inclusion Criteria

* Voluntary participation with signed informed consent
* Presence of symptoms consistent with carpal tunnel syndrome (CTS) (pain and/or paresthesia in the median nerve distribution), clinical signs (i.e., positive Tinel's and/or Phalen's test results), and electrodiagnostic findings (demonstrating mild to moderate CTS based on sensory or motor conduction studies of the median nerve)

Exclusion Criteria:

* Electrodiagnostic evidence of severe CTS
* Abnormal ulnar nerve conduction findings
* History of surgery for CTS
* History of physical therapy or injection for CTS within the past 6 months
* History of wrist fracture
* Presence of other conditions causing similar symptoms, such as polyneuropathy, cervical radiculopathy, ulnar neuropathy, brachial plexopathy, or thoracic outlet syndrome
* Central nervous system disorders (e.g., stroke, multiple sclerosis, Parkinson's disease)
* Pregnancy
* Presence of risk factors for CTS such as rheumatologic diseases, chronic kidney disease, diabetes mellitus, or hypothyroidism
* Malignancy
* Contraindications to rPMS (e.g., pacemaker, cochlear implant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | Baseline, three weeks after the final treatment session, and six weeks post-treatment.
  The Visual Analog Scale is a tool used to quantitatively assess pain intensity. It consists of a 10 cm horizontal line, with opposing descriptors at each end. The left end represents "no pain," and the right end represents "worst imaginable pain." Patients are asked to mark a point along the line that best represents the average level of pain they experience. The distance from the left endpoint to the point marked by the participant will be measured in centimeters and recorded as a VAS pain score.

SECONDARY OUTCOMES:
Grip and Pinch Strength Assessment | baseline, three weeks after the final treatment session, and six weeks post-treatment.
  Grip and pinch strength measurements are used to evaluate hand function and to quantitatively monitor progress throughout the treatment process. Grip strength is measured with the patient seated, shoulder adducted and neutrally rotated, elbow flexed at 90°, and the wrist in a neutral position. A Jamar dynamometer is used, and the average of three consecutive measurements is recorded. The same arm positioning is used for the pinch strength assessment. Three types of pinch are evaluated with a pinch gauge. Palmar pinch is assessed by bringing the thumb, index, and middle fingertips together. Lateral pinch is performed by pressing the distal phalanx of the thumb against the lateral surface of the middle phalanx of the index finger. Tip-to-tip pinch is evaluated by forming an "O" shape with the tips of the thumb and index finger. Each measurement is performed three times, and the average is recorded as kilograms (kg).
Boston Carpal Tunnel Questionnaire (BCTQ) | baseline, three weeks after the final treatment session, and six weeks post-treatment.
  The BCTQ is designed to evaluate symptom severity and functional status in patients with carpal tunnel syndrome. The questionnaire consists of two sections. The Symptom Severity Scale includes 11 items that evaluate the intensity, character, frequency, and duration of symptoms. Each item is rated on a scale from 1 (mildest) to 5 (most severe), and the final score is calculated as the arithmetic mean of all item scores. The Functional Status Scale comprises 8 items assessing the level of difficulty experienced in performing daily activities. Similar to the symptom scale, each item is scored between 1 and 5, and the average of these scores constitutes the final result. Higher scores in both sections indicate more severe symptoms and greater functional impairment.
SF-36 (Short Form-36 Health Survey Questionnaire) | baseline, three weeks after the final treatment session, and six weeks post-treatment.
  The SF-36 is a multidimensional questionnaire originally developed in the United States to evaluate general health status. The SF-36 consists of 36 items grouped into eight health domains, including physical functioning, role limitations due to physical and emotional problems, pain, general health perception, mental health, social functioning, and energy/fatigue.Each domain is scored on a 0-100 scale, where higher scores indicate better health status, lower scores reflect greater disability or poorer quality of life
Electrophysiological Evaluation | baseline, three weeks after the final treatment session, and six weeks post-treatment.
  All measurements will be performed at room temperature using the Keypoint®-Dantec EMG system available in our clinic. The patient will be positioned supine with the palm facing upward. For motor conduction studies, the active electrode will be placed over the abductor pollicis brevis muscle, and the reference electrode over the proximal phalanx of the thumb. Stimulation will be applied 8 cm proximally, and measurements will include distal motor latency (ms) and compound muscle action potential (CMAP, mV). For sensory conduction studies, the active electrode will be placed over the proximal phalanx of the index finger, and the reference electrode about 3-4 cm distally. Sensory conduction will be assessed orthodromically at the Digit 1-wrist, Digit 2-wrist, Palm-wrist, Digit 3-wrist, and Wrist-elbow segments.Measurements will include distal sensory latency (ms), sensory nerve action potential amplitude (SNAP, µV), and conduction velocity.
Ultrasonographic Measurement of Median Nerve Cross-Sectional Area | baseline, three weeks after the final treatment session, and six weeks post-treatment.
  The cross-sectional area of the median nerve will be assessed using an ultrasound (GE Healthcare Versana Premier) with a 7-12 MHz linear transducer. The forearm will be positioned in supination with the palm facing upward. At the level of the carpal tunnel, the area will be measured using manual tracing along the hyperechoic inner border of the nerve. The arithmetic mean of three consecutive measurements will be calculated and recorded in mm².

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Faculty of Medicine, Cebeci Hospital, Cebeci, Ankara, Mamak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No